CLINICAL TRIAL: NCT04143971
Title: Effects of Intermittent Fasting Compared to Continuous Calorie Restriction on Weight Loss & Plasma Lipids in Hypertriglyceridemic Overweight or Obese Subjects
Brief Title: Intermittent Fasting in Hypertriglyceridemic Overweight or Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University (Other)
Collaborators: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Nasrollahzadeh, Director, Shahid Beheshti University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 896
Record Dates: First submitted 2019-10-27; First posted 2019-10-30 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Hypertriglyceridemia; Overweight or Obesity
Keywords: intermittent fasting; hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia; Overweight; Obesity; Intermittent Fasting | interventions — Caloric Restriction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continiuous Low calorie diets (Placebo Comparator): Low calorie diet with daily calorie restriction
  Interventions: Other: low calorie diet
- Intermittent Fasting (Active Comparator): Intermittent fasting every other day, in which daily calorie intake will be up to 30% of required calorie.
  Interventions: Other: intermittent fasting diet

INTERVENTIONS:
Other: intermittent fasting diet — intermittent fasting diet
  Arms: Intermittent Fasting
Other: low calorie diet — continuous low calorie diet
  Arms: Continiuous Low calorie diets

SUMMARY:
some studies have shown similar effects of intermittent fasting and continuous caloric restriction on body weight and plasma lipid profile, but there is still a wide controversy. Therefore,due to limited human studies and the lack of a study on hypertriglyceridemic patients, the present study aimed to determine the effects of using low-calorie diets in comparison with continuous caloric restriction on weight loss and plasma lipid profile in obese or overweight hypertriglyceridemic patients.

DETAILED DESCRIPTION:
a randomized clinical trial will be conducted in National Nutrition and Food Technology Research Institute, Tehran, Iran. after the review of inclusion and exclusion criteria, a written consent form will be completed. the participants will be 90 hypertriglyceridemic patients aged between 18-60. half of the participants will be under intermittent low-calorie diet which they will have 3 alternate days in the week eating only 30% of their total energy requirement and on the other days of the week they receive a total calorie of 100% of their energy requirement , therefore there will be a total of -210% TEE reduction in their received energy in the week. the other group will be under continuous calorie restriction meaning on all the days of the week they will be eating 70% of their total energy requirement resulting in a total of -210% TEE reduction in their received energy in the week. both groups will receive 3 consultation sessions with a nutritionist, also to prevent any deficiency, multi-vitamin-mineral supplements will be given to both groups participants.

ELIGIBILITY:
Inclusion Criteria:

* hypertriglyceridemic : TG>150 mg/dL
* BMI>24.9
* age 18-60
* non-smoker
* haven't been under any diet at least 3 months before participating in the study
* not starting any new exercise program or changing the previous exercise while in the study

Exclusion Criteria:

* chronic kidney disease stage 3-5
* consuming Insulin or Insulin-inducing drugs.
* consuming triglycerides lowering drugs or Omega 3
* a history of cholecystitis
* Heart arrhythmia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Weight loss | at 8 weeks
  Mean weight change of participants (kg) after 8 weeks of diets

SECONDARY OUTCOMES:
Plasma Triglycerides | at 8 weeks
  Mean change in plasma triglycerides of participants after 8 weeks of diets

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Unit, National Nutrition and Food Technology Research Institute, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maroofi M, Nasrollahzadeh J. Effect of intermittent versus continuous calorie restriction on body weight and cardiometabolic risk markers in subjects with overweight or obesity and mild-to-moderate hypertriglyceridemia: a randomized trial. Lipids Health Dis. 2020 Oct 7;19(1):216. doi: 10.1186/s12944-020-01399-0. PMID 33028352